CLINICAL TRIAL: NCT06873698
Title: A Pilot Randomized Controlled Trial (RCT) of Neurobehavioral Therapy (NBT) Vs Standard Medical Care (SMC) for Functional Neurological Disorder (FND)
Brief Title: Pilot Neurobehavioral Therapy for Functional Neurological Disorder
Acronym: NBT for mFND
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Principal Investigator, W. Curt LaFrance Jr., MD, MPH, Professor / Principal Investigator, Rhode Island Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2136841
Record Dates: First submitted 2025-03-07; First posted 2025-03-13 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Functional Neurological Disorder
Keywords: mFND; Conversion Disorder; Functional Neurologic Disorder; Neurobehavioral Therapy; FND; Psychogenic Movement Disorder; Psychotherapy; motor functional neurological disorder; functional motor disorder
MeSH Terms: conditions — Conversion Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Neuro-Behavioral Therapy (Experimental): Participants will receive neuro-behavioral therapy (NBT), in individual, weekly, one-hour appointments, using the 12 session, "Taking Control of Your Functional Movements: Workbook", over the course of 12 to 18 weeks.
  Before each appointment, participants will complete worksheets/questions in one chapter that will be discussed during the weekly virtual appointment. Video appointments will be completed using an encrypted healthcare weblink and will be digitally recorded for review to ensure therapy adherence and competence. Participants randomized to the NBT arm will also participate in 5 in-person visits for exam documentation.
  Interventions: Behavioral: Neuro-behavioral Therapy
- Standard Medical Care (Active Comparator): If randomized to this treatment arm, participants will continue to follow up with their clinicians while receiving standard medical care (SMC) and without receiving the study intervention. Research staff will ask about what care participants are receiving when they meet with staff. Subjects randomized to the SMC arm will participate in 5 in-person visits for exam and SMC documentation.
  Interventions: Other: Standard Medical Care (SMC)

INTERVENTIONS:
Behavioral: Neuro-behavioral Therapy — Neuro-behavioral therapy (NBT) is an evidence-based, multi-modality, time-limited, whole-person therapy, delivered in one hour, weekly, individual appointments. NBT has been used to treat epilepsy, nonepileptic (functional) seizures, and motor functional neurological disorder (mFND).
  Other Names: Taking Control of Your Functional Motor Disorder Workbook
  Arms: Neuro-Behavioral Therapy
Other: Standard Medical Care (SMC) — Standard Medical Care (SMC) involves the routine care received by the participant. SMC may include any of the following evaluation and followup appointments with neurology, physiatry, psychiatry, psychology, mental health, rehabilitation (e.g., Physical Therapy, Occupational Therapy, Speech and Language Therapy), primary care, among other specialists.
  Arms: Standard Medical Care

SUMMARY:
The goal of this pilot randomized clinical trial is to learn if Neurobehavioral Therapy (NBT) works to treat motor functional neurological disorder (mFND) (also referred to as functional motor disorder).

The main questions it aims to answer are:

* Does NBT lower mFND symptoms?
* Does NBT lower common co-occurring symptoms and improve functioning?

Researchers will compare NBT to standard medical care (SMC).

Participants will be randomized to receive either:

* 12 weekly sessions of NBT, along with their SMC,
* or continue receiving their SMC as provided by their treating clinicians.
* all participants. regardless of group assignment, will complete a total of five in-clinic visits at the following time points: Baseline, 6 weeks, 12 weeks, 8 Months and 12 Months for self-report surveys to assess functional status, quality of life and mFND symptoms.

DETAILED DESCRIPTION:
The study aims to enroll 40 participants at Rhode Island Hospital. 20 participants with Motor Functional Neurological Disorder (mFND) will be randomized to Neurobehavioral Therapy (Group 1) and 20 participants with mFND to Standard Medical Care (Group 2). Those randomized to neurobehavioral therapy will be asked to complete treatment sessions over the course of 12 to 18 weeks. Those in the standard medical care arm will continue to receive their routine care with their clinicians.

All participants regardless of group assignment, will complete a total of five in-person clinic visits at the following time points: Baseline, 6 weeks, 12 weeks, 8 Months and 12 Months. These visits will include the completion of interview questions and self-report surveys that will assess functional status, quality of life and mFND symptoms.

Please see the "Arms and Interventions" section to see a more detailed description of each group/arm.

The goal of this Clinical Trial is to investigate the feasibility and efficacy of Neuro-Behavioral Therapy in Individuals aged 18 to 70 diagnosed with Motor Functional Neurologic Disorder. The main questions this study aims to answer are:

Aim 1: Examine the feasibility, acceptability, and practicality of manualized Neuro-Behavioral Therapy (NBT) in Functional Neurological Disorder (FND).

Hypothesis 1: Manualized NBT will demonstrate feasibility through acceptability and practicality, defined as ≥80% of participants enrolling in the study will participate in the study measures (acceptability) and complete the entire study protocol (practicality), respectively.

Aim 2: Examine the preliminary effectiveness of manualized NBT in improving health-related quality of life and reducing the severity and disability of mFNDs, as measured by the SF-36 and PMDRS/S-FMDRS (primary outcome), respectively.

Hypothesis 2: NBT will show improvements in SF-36 scores and reductions in PMDRS scores. We will evaluate this by conducting a preliminary examination of the manualized NBT intervention, with a focus on interpreting effect sizes. We will also gather key statistics needed to inform a fully powered clinical trial, such as the standard deviation and pre-post correlation of the SF-36 and PMDRS.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with Motor Functional Neurological Disorder (mFND)
* Individuals aged 18-70 years
* At least 1 mFND symptom during the year prior to enrollment

Exclusion Criteria:

* Current or past year self-injurious behavior
* Current suicidality (PHQ-9 question 9 rated as 1 or above)
* Current or past year psychosis
* Pending litigation or current application for long term disability
* Active substance or alcohol use disorders (dependence), at the discretion of the investigator if they preclude participation in the study
* Serious illness requiring systemic treatment or hospitalization; the participant either completes therapy or is clinically stable on therapy, for at least 30 days prior to study entry
* Inability to fill out the self-report surveys
* Inability or unwillingness to participate in NBT and assigned homework
* Currently enrolled in NBT aimed at mFND

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-09-25 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
SF-36 Health Survey (SF-36) | Baseline, Week 6, Week 12, 8 Months and 12 Months
  The SF-36 is a 36-item self-report measure that assess 8 domains: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions.
Psychogenic Movement Disorders Rating Scale (PMDRS) | Baseline, Week 6, Week 12, 8 Months and 12 Months
  The PMDRS is a clinical assessment tool designed to measure the severity and characteristics of abnormal movements associated with psychogenic movement disorders (also called functional movement disorders), including details like the type of movement, affected body regions, duration, and functional impact of the symptoms, allowing clinicians to track changes over time and evaluate treatment efficacy.
Simplified Functional Movement Disorders Rating Scale (S-FMDRS) | Baseline, Week 6, Week 12, 8 Months and 12 Months
  The S-FMDRS is a clinical tool used to assess the severity of functional movement disorders (FMDs) by evaluating the presence and intensity of abnormal movements in different body regions, including gait and speech.

SECONDARY OUTCOMES:
Generalized Anxiety Disorder (GAD-7) | Baseline, Week 6, Week 12, 8 Months and 12 Months
  The GAD-7 is a 7 item self-report measure that assesses Anxiety severity from "0" (not at all) to "3" (nearly every day) on each question. The highest possible score is "21", relating to the highest severity of Generalized Anxiety Disorder.
Patient Health Questionnaire (PHQ-9) | Baseline, Week 6, Week 12, 8 Months and 12 Months
  The PHQ-9 is a 9-item self-report measure instrument that assesses the severity of Depression on a scale from "0" (not at all) to "3" (nearly every day). The maximum score is 27.
Patient Health Questionnaire (PHQ-15) | Baseline, Week 6, Week 12, 8 Months and 12 Months
  The PHQ-15 is a 15-item self-report measure instrument that assesses the presence and severity of somatic symptoms on a scale from "0" (not bothered at all) to "2" (bothered a lot). The maximum score is 30.
Posttraumatic Scale Checklist-5 (PCL-5) | Baseline, Week 6, Week 12, 8 Months and 12 Months
  The PCL-5 is a 20-item self-report measure that assesses the presence and severity of PTSD symptoms.
Global Assessment of Functioning (GAF) | Baseline, Week 6, Week 12, 8 Months and 12 Months
  This GAF rating scale ranges from 0 (worst) to 100 (best) and is used for evaluating the overall functioning and symptoms of an individual during a specified time period on a continuum from psychological or psychiatric sickness to health.
Clinical Global Impressions - Severity (CGI-S) | Baseline, Week 6, Week 12, 8 Months and 12 Months
  The CGI-S is the first item of a two-item global rating scale, where each item is on a 7 point scale ranging from normal ("1") to among the most extremely ill patients ("7"). A higher score relates to a higher severity of illness.
Clinical Global Impressions - Improvement (CGI-I) | Baseline, Week 6, Week 12, 8 Months and 12 Months
  The CGI-I is the second item of a two item global rating scale, where each item is on a 7 point scale ranging from very much improved ("1") to very much worse ("7"). A lower score represents a higher improvement.
World Health Organization: Quality of Life - BREF (WHOQOL-BREF) | Baseline, Week 6, Week 12, 8 Months and 12 Months
  This is a 27-item self-report scale to evaluate Quality of Life. The lowest possible score is 0 and the highest possible score is 100, reflecting a better quality of life.
Patient Reported Outcome Measurement Information System (PROMIS) 29+2 v2.1 | Baseline, Week 6, Week 12, 8 Months and 12 Months
  The PROMIS 29+2 v.2.1 is a 29 item self-report measure that assesses seven key health domains: physical function, anxiety, depression, fatigue, sleep disturbance, ability to participate in social roles and activities, and pain interference.
Multidimensional Health Locus of Control (MHLC-C) | Baseline, Week 6, Week 12, 8 Months and 12 Months
  The MHLC-C is a 18 item self-report measure that assesses how individuals view control over their health when dealing with a specific condition. It looks at three beliefs: (1) whether individuals feel in control of their health (Internal), (2) whether individuals rely on doctors or others (Powerful Others), or (3) whether individuals think health is mostly luck or chance (Chance). This survey helps to understand how these three beliefs may influence how individuals manage their condition.
Traumatic Life Events Questionnaire (TLEQ) | Baseline
  The TLEQ is a 17-item self-report measure that assesses individuals experiences with potentially traumatic events, such as accidents, natural disasters, or violence. The TLEQ helps to identify whether someone has been exposed to trauma, how often these events have occurred and how impact or distressing these events were on ones well-being.
Montreal Cognitive Assessment (MoCA) | Baseline, Week 12, and 12 Months
  The MoCA is a 30 item assessment tool used to detect mild cognitive impairment by evaluating various cognitive domains like memory, attention, language, visuospatial abilities, executive function, and orientation. The scale has a total possible score of 30 points, where a score of 26 or higher is typically considered normal while a lower score may indicate potential cognitive impairment.

OTHER OUTCOMES:
Abnormal Movement Log | Baseline, [Weekly - NBT Arm Only], Week 6, Week 12, 8 Months and 12 Months
  The Abnormal Movements Log is a daily diary to track unusual movements over the course of a week. Each day, individuals will record a series of details in relation to their mFND such as the number, duration, time, body parts affected, type of movement, severity (mild, moderate, severe), triggers, warning signs, what helps, and how it impacts themselves and others. The Principal Investigator will review the movement logs during study visits to better understand ones symptoms and how impactful they are one ones day. It's a simple tool aimed to identify patterns and improve care.
Status Survey | Baseline, Week 6, Week 12, 8 Months and 12 Months
  The Status Survey is a 17 item self report measure that assesses research participants experience with motor Functional Neurological Disorder (FND) through the duration of the trial. The survey asks about current symptoms, emergency room visits, medications (for movement, anxiety, or depression), new therapies, and any new or worsening symptoms. It also includes questions about individuals daily life, such as work, disability status, driving, and overall quality of life over the past four weeks. The goal is to gather updates on how individuals are managing FND and its impact on ones well-being.

CONTACTS AND LOCATIONS:
Overall Officials: W. Curt LaFrance Jr, MD, MPH, Principal Investigator — Brown University Health; Emily Weisbach, MD, Study Chair — Brown University Health
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data used in the current study will be available after termination of the embargo period or upon reasonable request from the authors with regulatory approval.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available after termination of the embargo period until IRB closure.
Access Criteria: Data will be made available to authors with regulatory approval upon reasonable request to the study Principal Investigator.

REFERENCES:
- [Background] LaFrance WC Jr, Tedesco R, Baird GL, Wincze J, Tocco K, Anderson J. Clinician-rated outcomes of patients with functional neurological disorders treated in an outpatient clinic. Seizure. 2023 Apr;107:21-27. doi: 10.1016/j.seizure.2023.03.005. Epub 2023 Mar 12. PMID 36933399